CLINICAL TRIAL: NCT04863170
Title: Cross Cultural Adaptation and Validation of Chilean Version of Orthognathic Quality of Life Questionnaire (OQLQ)
Brief Title: Cross Cultural Adaptation and Validation of Orthognathic Quality of Life Questionnaire (OQLQ)
Status: Completed | Type: Observational
Sponsor: Hospital Carlos Van Buren (Other)
Collaborators: Universidad de La Frontera (Other); University of Chile (Other); Pontificia Universidad Catolica de Valparaiso (Other); Hospital San Borja-Arriaran (Other); Universidad de Valparaiso (Other); Hospital del Mar Research Institute (IMIM) (Other)
Responsible Party: Sponsor
Other Study IDs: ORD 2436 / 30-11-18
Record Dates: First submitted 2021-04-02; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Health-related Quality of Life; Dentofacial Deformities
Keywords: Health-related quality of life; Orthognathic surgery; Dentofacial deformities
MeSH Terms: conditions — Dentofacial Deformities | interventions — Orthognathic Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: orthognathic surgery — surgical intervention of the maxilla and / or mandible that includes orthodontic treatment before and after surgery

SUMMARY:
The aim of this study was to develop a Spanish version of the Orthognathic Quality of Life Questionnaire (OQLQ) that is conceptually equivalent to the original questionnaire, as well as acceptable, reliable, valid, and responsive for use in Chilean patients with dentofacial deformities.The cross cultural adaptation process was carried out according to the recommended standard methodology with direct and back-translation.

DETAILED DESCRIPTION:
A prospective longitudinal multicenter study of adult patients diagnosed with dentofacial deformity was carried out, self-administrating OQLQ, OHIP-14 (Oral Health Impact Profile), and SF-36 (Short Form 36 Health Survey) during the presurgery visit in order to examine construct validity. To evaluate reproducibility, questionnaires were re-administered 4 weeks later to subjects with a stable dental condition. Responsiveness was assessed among subjects followed up until 3 months after surgery and finally changes in health-related quality of life was assessed comparing baseline pre-surgery to 3 and 6 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients over 18 years old with dentofacial deformity.

Exclusion Criteria:

* Patients with congenital abnormalities such as craniofacial syndrome or cleft lip/palate and sequels due to maxillofacial trauma were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients over 18 years old with dentofacial deformity Class II or III in orthodontic-surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Metric properties of Orthognathic Quality of Life Questionnaire (OQLQ): Reliability | 4 weeks follow-up
  To measure this metric property, internal consistency and test-retest reproducibility were assessed. The orthognathic quality of life questionnaire (OQLQ) was applied twice, with four weeks between tests.
  To assess reliability, the internal consistency was estimated by the Cronbach alpha coefficient, and the test-retest reproducibility was estimated by the intraclass correlation coefficient.
  The orthognathic quality of life questionnaire is a condition specific instrument for assessment oral health quality of life in dentofacial deformities patients 22 ítems values: min = 0 / max = 88 higher scores mean a worse outcome
Metric properties of Orthognathic Quality of Life Questionnaire (OQLQ): Validity | baseline
  Validity refers to the degree to which the instrument measures what it purports to measure.
  Construct validity was evaluated analyzing the hypothesized relationships between scores by calculating the Spearman correlation coefficients.
  The orthognathic quality of life questionnaire is a condition specific instrument for assessment oral health quality of life in dentofacial deformities patients 22 ítems values: min = 0 / max = 88 higher scores mean a worse outcome
Metric properties of Orthognathic Quality of Life Questionnaire (OQLQ): Responsiveness to change | baseline - 3 months follow-up
  Responsiveness refers to an instrument's ability to detect change. To evaluate responsiveness of the orthognathic quality of life questionnaire (OQLQ) we applied twice: first one week before surgery (T1), and then three months after surgery (T2) To evaluate responsiveness, a paired t-test was used to assess the score changes in patients undergoing orthognathic surgery. The magnitude of the change was evaluated calculating the standardized response mean.
  The orthognathic quality of life questionnaire is a condition specific instrument for assessment oral health quality of life in dentofacial deformities patients 22 ítems values: min = 0 / max = 88 higher scores mean a worse outcome
changes in oral health related quality of life after orthognathic surgery assessed with Orthognathic Quality of Life Questionnaire (OQLQ) | baseline to 3 and 6 months follow-up
  Orthognathic quality of life questionnaire (OQLQ) was applied at 3 times: baseline, one week before surgery (T1), three months after surgery (T2) and 6 months after surgery (T3).
  A paired t-test was used to assess the mean (SD) changes in patients undergoing orthognathic surgery. The magnitude of the change was evaluated calculating the standardized response mean (SRM).
  The orthognathic quality of life questionnaire is a condition specific instrument for assessment oral health quality of life in dentofacial deformities patients 22 ítems values: min = 0 / max = 88 higher scores mean a worse outcome
changes in oral health related quality of life after orthognathic surgery assessed with Short form Oral Health Impact Profile (OHIP-14) | baseline to 3 and 6 months follow-up
  Short form Oral Health Impact Profile (OHIP-14) was applied at 3 times: baseline, one week before surgery (T1), three months after surgery (T2) and 6 months after surgery (T3).
  A paired t-test was used to assess the mean (SD) changes in patients undergoing orthognathic surgery. The magnitude of the change was evaluated calculating the standardized response mean (SRM).
  The Short Form Oral Health Impact Profile (OHIP-14) is an instrument for assessment oral health-related quality of life.
  14 ítems values: min = 0 / max = 56 higher scores mean a worse outcome
changes in health related quality of life after orthognathic surgery assessed with Short Form Health Survey (SF-36) | baseline to 3 and 6 months follow-up
  The Short Form Health Survey (SF-36) was applied at 3 times: baseline, one week before surgery (T1), three months after surgery (T2) and 6 months after surgery (T3).
  A paired t-test was used to assess the mean (SD) changes in patients undergoing orthognathic surgery. The magnitude of the change was evaluated calculating the standardized response mean (SRM).
  The Short Form Health Survey (SF-36) is a generic health-related quality of life questionnaire 36 ítems in addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
  higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Duarte, Principal Investigator — Hospital Carlos Van Buren
Locations (1):
- Valentina Duarte, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No